CLINICAL TRIAL: NCT07315724
Title: The Efficacy of a Technology-Assisted Block Training Program on Cognitive Function, Hand Dexterity, and Grip Strength in Community-Dwelling Older Adults: A Mixed-Methods Research
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chia Jung Hsieh, Ph.D., RN, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FJU-IRB NO:C113099
Record Dates: First submitted 2025-11-16; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Community-Dwelling Older Adults; Aging; Cognitive Decline; Hand Dexterity; Muscle Strength
Keywords: Technology-assisted block training program; Block-building activities; Cognitive function; Hand dexterity; Grip strength; Older adults; Mental rotation; Mixed-methods research; Spatial cognition; Quality of life
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Single Group, pre-post test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single group (Experimental): This intervention arm involves a weekly 2-hour building block course that incorporates mental rotation training components. Participants will engage in structured building block activities designed to enhance spatial reasoning abilities, with specific lesson plans focused on developing mental rotation skills through hands-on construction and manipulation of three-dimensional objects.
  Interventions: Behavioral: Technology-Assisted Block Training Program

INTERVENTIONS:
Behavioral: Technology-Assisted Block Training Program — This study, drawing on the theories proposed by Aguilar Ramirez et al. (2022) and Shepard and Metzler (1971), developed a mental rotation application and a corresponding block-building lesson plan. Participants then engaged in individual block-building activities, guided by the lesson plan, to train their spatial reasoning skills. Finally, the developed APP was used for mental rotation training, and its suitability and feasibility were rigorously validated through expert review and a pilot study. a. Mental Rotation Virtual Reality APP: The APP's content was validated by interdisciplinary experts (including gerontology, activity planning, cognitive training, and information technology) to ensure its appropriateness and feasibility. The APP incorporates technology-assisted elements, such as real-time feedback and personalized difficulty adjustment for the mental rotation exercises, to enhance training effectiveness and participant motivation. Furthermore, the built-in "Creative Showcase"

SUMMARY:
Block-building activities represent a promising tool for enhancing cognitive and hand function in older adults. When integrated with technological support, they offer personalized training advantages; however, their comprehensive effectiveness requires empirical validation. This study aimed to develop and evaluate a "Technology-Assisted Block Training Program" to explore its effects on cognitive function, hand grip strength, dexterity, and quality of life among community-dwelling older adults, while examining participants' subjective experiences.

DETAILED DESCRIPTION:
In response to the aging population trend, developing evidence-based care programs for older adults has become increasingly necessary. To delay functional decline in individuals, intervention programs that combine cognitive and motor training are gaining greater attention. Manual activities such as block-building can effectively improve working memory and processing abilities. However, traditional block training and cognitive training often struggle to maintain participants' motivation and sustained engagement due to monotonous content. Therefore, technology-assisted block training has emerged as a solution, providing real-time feedback, personalized difficulty adjustment, and multi-sensory stimulation to effectively overcome the limitations of traditional training approaches and enhance participant motivation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 65 and older
2. Mentally alert and able to communicate
3. Willing to participate in this study

Exclusion Criteria:

1. Diagnosed with dementia by a physician
2. Severe sensory or communication impairment
3. Hand function impairment that prevents manipulation of building blocks

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function - Montreal Cognitive Assessment (MoCA) | Time Frame: Baseline, pre-intervention
  Description:
  The MoCA is a 30-point cognitive screening tool with established reliability in older adults. Higher scores indicate better cognitive function.
  Unit of Measure:
  Points on a 30-point scale
Spatial Cognition - Mental Rotation Test | Baseline , pre-intervention
  Description:
  The Mental Rotation Test assesses spatial cognition. Higher numbers of correct responses indicate better mental rotation ability.
  Unit of Measure:
  Number of correct responses
Hand Grip Strength - Jamar Hydraulic Hand Dynamometer | Baseline ,pre-intervention
  Description:
  Grip strength of each hand is measured using the Jamar dynamometer. Three trials per hand will be averaged. Higher values indicate greater grip strength.
  Unit of Measure:
  Kilograms (kg)
Hand Dexterity - Purdue Pegboard Test | Baseline ,pre-intervention
  Description:
  The Purdue Pegboard Test assesses fine motor skills and dexterity of the hands and fingers. The score reflects the number of pegs correctly placed in the allotted time.
  Unit of Measure:
  Number of pegs placed
Well-Being - WHO-5 Well-Being Index | Baseline , pre-intervention
  Description:
  The WHO-5 consists of five items rated on a 25-point scale. Higher scores indicate better well-being and quality of life.
  Unit of Measure:
  Points on a 25-point scale
System Usability - System Usability Scale (SUS) | Baseline , pre-intervention
  Description:
  The SUS assesses usability, learnability, and satisfaction with technology-based systems. Scores range from 0 to 100; higher scores indicate better usability.
  Unit of Measure:
  Score on a 0-100 scale

SECONDARY OUTCOMES:
Cognitive Function - Montreal Cognitive Assessment (MoCA) | Immediately After the 4-week Intervention
  Description:
  The MoCA is a 30-point cognitive screening tool with established reliability in older adults. Higher scores indicate better cognitive function.
  Unit of Measure:
  Points on a 30-point scale
Spatial Cognition - Mental Rotation Test | Immediately After the 4-week Intervention
  Description:
  The Mental Rotation Test assesses spatial cognition. Higher numbers of correct responses indicate better mental rotation ability.
  Unit of Measure:
  Number of correct responses
Hand Grip Strength - Jamar Hydraulic Hand Dynamometer | Immediately After the 4-week Intervention
  Description:
  Grip strength of each hand is measured using the Jamar dynamometer. Three trials per hand will be averaged. Higher values indicate greater grip strength.
  Unit of Measure:
  Kilograms (kg)
Hand Dexterity - Purdue Pegboard Test | Immediately After the 4-week Intervention
  Description:
  The Purdue Pegboard Test assesses fine motor skills and dexterity of the hands and fingers. The score reflects the number of pegs correctly placed in the allotted time.
  Unit of Measure:
  Number of pegs placed
Well-Being - WHO-5 Well-Being Index | Immediately After the 4-week Intervention
  Description:
  The WHO-5 consists of five items rated on a 25-point scale. Higher scores indicate better well-being and quality of life.
  Unit of Measure:
  Points on a 25-point scale
System Usability - System Usability Scale (SUS) | Immediately After the 4-week Intervention
  Description:
  The SUS assesses usability, learnability, and satisfaction with technology-based systems. Scores range from 0 to 100; higher scores indicate better usability.
  Unit of Measure:
  Score on a 0-100 scale

CONTACTS AND LOCATIONS:
Locations (1):
- Xindong Community Activity Center, Yilan City, Yilan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT07315724/Prot_SAP_ICF_000.pdf